CLINICAL TRIAL: NCT01770041
Title: Observational Study Assessing Cytochrome P450 Dependant Paracetamol Metabolites Following Liver Resection.
Brief Title: Paracetamol Metabolism After Liver Surgery
Acronym: PETALS
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 12/SS/0222
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Liver Resection; Paracetamol Administration
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Liver resection group: Patients undergoing liver resection and receiving paracetamol (observation of routine administration)
  Interventions: Other: Paracetamol (observation of routine administration)

INTERVENTIONS:
Other: Paracetamol (observation of routine administration) — Normal administration of paracetamol as prescribed by operating surgeon
  Other Names: Acetaminophen

SUMMARY:
This observational study will assess the metabolic pathways of paracetamol that are utilised after liver resection.

DETAILED DESCRIPTION:
Paracetamol is normally metabolised by the glucuronidation and sulfation of paracetamol to non toxic end products. If paracetamol is administered in supra-therapeutic doses this pathway becomes saturated and an alternative pathway is utilised. This results in a toxic metabolite called N-acetyl-p-benzoquinone imine (NAPQI). If NAPQI is not metabolised by glutathione to cysteine and mercapturic acid, then NAPQI bind to hepatic cells resulting in necrosis and hepatotoxicity.

Therefore the investigators plan to measure the levels of the paracetamol metabolites in patient undergoing liver resection.

Patients will undergo liver resection according to their onco-surgical requirements. As part of the normal post operative care they will receive 1g paracetamol every six hours unless stated otherwise by the operating surgeon. Urinary samples will be taken for the first 4 post operative days and used for analysis of the urinary paracetamol metabolite levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver surgery

Exclusion Criteria:

* Contra-indication to paracetamol
* Inability to give written, informed consent.
* Jaundice (Bilirubin > 100 μmol/L).
* Liver resection combined with secondary surgical procedure.
* Age < 18 years.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with benign or malignant liver tumours that have been deemed by the hepatobiliary multi-disciplinary team meetiong as requiring surgical intervention.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Urinary cysteine | Post operative days 1-4

SECONDARY OUTCOMES:
mercapturic acid | post operative days 1-4
Glutathione | day of surgery and post operative days 1 and 3
Paracetamol level | day of surgery and post operative days 1 and 3

OTHER OUTCOMES:
Glucuronamide | Post-operative days 1-4
Sulphate | Post-operative days 1-4
5-oxoproline | Post-operative days 1-4
Complications | Day of surgery and post-operative days 1-30
Post-operative blood tests (FBC, U&E, LFTs, Coag) | Post-operative dyas 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Hughes, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom